CLINICAL TRIAL: NCT03389919
Title: EFFECTIVENESS AND SAFETY OF INTRAOSSEOUS ADMINISTRATION OF MESENCHYMAL STORMAL CELLS FOR PRIMARY GRAFT FAILURE AFTER ALLOGENEIC STEM CELL TRANSPLANTATION
Brief Title: Intraosseous Administration of Mesenchymal Stromal Cells for Patients With Graft Failure After Allo-HSCT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Research Center for Hematology, Russia (Network)
Responsible Party: Principal Investigator, Elena N.Parovichnikova, Head of BMT department, National Research Center for Hematology, Russia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BM-MSC-01
Record Dates: First submitted 2017-12-27; First posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Mesenchymal Stem Cell Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: MSC administration (intraosseal) — MSCs will be administered under local anesthesia to the iliac crests after receiving informed consent from the patient.

SUMMARY:
Multipotent mesenchymal stromal cells (MSCs) participate in the formation of bone marrow niches for hematopoietic stem cells. Donor MSCs can serve as a source of recovery for niches in patients with graft failure (GF) after allogeneic bone marrow (BM) transplantation. Since only few MSCs reach the BM after intravenous injection, MSCs were implanted into the iliac spine. Preliminary results suggest that MSCs participate in the restoration of niches for donor hematopoietic cells or have an immunomodulatory effect, preventing repeated rejection of the graft. Perhaps intraosseous implantation of MSCs contributes to the success of the second transplantation of hematopoietic stem cells and patient survival.

ELIGIBILITY:
Inclusion Criteria:

* All patients with primary graft failure after allo-HSCT
* Available MSC for this patient

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Engraftment | 28-day
  Engraftment

CONTACTS AND LOCATIONS:
Locations (1):
- BMT department, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided